CLINICAL TRIAL: NCT00350350
Title: Multicenter, Controlled Parallel Groups Trial to Evaluate the Efficacy, Safety and Acceptability of OGT Oromucosal Spray Versus a Saliva Substitute in the Treatment of Xerostomia in Geriatrics
Brief Title: OGT Spray in the Management of Xerostomia in the Elderly
Status: Completed | Type: Observational
Sponsor: Laboratoires CARILENE (Industry)
Collaborators: Eurofins Dermscan Pharmascan (Industry)
Responsible Party: Sponsor
Other Study IDs: CARILENE LABORATORY
Record Dates: First submitted 2006-07-06; First posted 2006-07-10 (Estimated); Last update posted 2012-04-23 (Estimated); Status verified 2006-07

CONDITIONS: XEROSTOMIA
Keywords: XEROSTOMIA; MOUTH DRYNESS; ELDERLY; ORAL LUBRICANT
MeSH Terms: conditions — Xerostomia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- elderly people: elderly people over 70 years residents of old's people homes with symptoms of dry mouth
  Interventions: Device: oxygenated oil; Device: medical device. Spray containing essentially oxygenated oil

INTERVENTIONS:
Device: oxygenated oil — oxygenated oil in spray versus product reference (artificial saliva) dosage : one to two spray 5 times a day
  Other Names: artificial saliva
Device: medical device. Spray containing essentially oxygenated oil — protective oral spray containing :
  * 94.4% of oxygenated oil
  * Silicium dioxide
  * aspartame artificial flavoring
  Other Names: artificial saliva

SUMMARY:
The primary objective of the trial is to evaluate the efficacy, safety and clinical acceptability of OGT oromucosal spray in the relief of symptoms and signs of xerostomia in comparison with a saliva substitute (European Medical Device).

DETAILED DESCRIPTION:
Xerostomia is excessive dryness of the mouth. It is due to insufficient (hyposialism) or inexistent (asialia) saliva secretion.

There are many causes. Transitory xerostomia may occur in the presence of anxiety (stage fright, fear or dehydration). Prolonged xerostomia is most often related to a systemic disease, certain medicines or to radiotherapy of the head or neck.

Xerostomia is often accompanied by buccal symptoms and signs such as impaired sense of taste, fetid breath and mouth ulcers, and it disturbs functions such as speech, chewing and swallowing. Because of reduced salivary secretion, there is disturbance of the microbial colonization of the buccal cavity, increased demineralization and decreased remineralization of the teeth, impaired retention of dentures, dehydration of the mucosa and reduced lubrication of the buccal mucosa. These complications may take the form of dental caries, candidiasis, atrophy and feelings of burning of the mucosa, difficulty retaining dentures, impaired speech and swallowing and impression of decreased or impaired sense of taste. Xerostomia has significant harmful effects on the buccal cavity and on the quality of life of patients.

Xerostomia prevalence rates of the order of 18-61% have been reported in the elderly. These rates are generally higher in women that in men and increase with age. They are also higher in populations in institutions and in those taking multiple medications. Wearing a denture, stress and other psychological factors have also been suggested as factors increasing risk or or worsening xerostomia.

Treatments of xerostomia are saliva substitutes and saliva stimulants.

OGT Spray is neither a substitute nor stimulant of saliva.

OGT Spray is a solution for oromucosal spray which has lubricant and protective actions.

The aim of the study was to demonstrate that OGT Spray (oral lubricant) was effective in the subjective relief of dry mouth symptoms and objective signs of dry mouth in elderly.

ELIGIBILITY:
Inclusion Criteria:

* male or female, institutionalized and at least 70 years of age
* with a diagnosis of xerostomia confirmed objectively by the saliva absorption test
* having stopped all palliative treatment for xerostomia
* legally capable of giving consent
* capable and agreeing to participate in the study and capable and accepting to answer study questionnaires in accordance with the terms of the French Huriet Act on clinical trials,
* remaining in the establishment throughout the study period

Exclusion Criteria:

* Concomitant treatments incompatible with the trial, especially alcoholic solutions
* buccal fungal infection
* systemic infection or current dental care
* current participation in other clinical trials
* allergy or known intolerance to one of the constituents of the trial products
* treatment with atropine
* presence of active life-threatening disease

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: elderly population at least 70 years old residents of old's people homes
Sampling Method: Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2003-10; Primary Completion 2004-11 (Actual); Study Completion 2004-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michel MS SALOM, Gerontologis, Principal Investigator — Clinique Leopold Bellan 78200 Magnanville, France
Locations (1):
- clinique Léopold Bellan, Magnanville, Yvelines, France

REFERENCES:
- [Background] Fox PC. Management of dry mouth. Dent Clin North Am. 1997 Oct;41(4):863-75. PMID 9344281